CLINICAL TRIAL: NCT06234462
Title: Feasibility Study of Amantadine for Cognitive Dysfunction in Patients With Long-Covid: A Pilot Randomized Control Trial
Brief Title: A Study of Amantadine for Cognitive Dysfunction in Patients With Long-Covid
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: challenges with recruitment
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Amy Mathews, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2023-0234
Record Dates: First submitted 2024-01-08; First posted 2024-01-31 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Long COVID; Post-Acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Amantadine; Restraint, Physical; Speech Therapy; Dosage Forms; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Participants in this arm will receive current standard of care for PASC symptoms which may include: PT, OT, SLP, provider counseling, and/or pharmacologic interventions for targeted symptom management.
  Interventions: Other: Physical, Occupational, Speech Therapy; Other: Provider Counseling; Other: Medications for symptoms management
- Standard of Care + Amantadine (Experimental): Participants in this arm will review standard of care and amantadine.
  Interventions: Drug: Amantadine; Other: Physical, Occupational, Speech Therapy; Other: Provider Counseling; Other: Medications for symptoms management

INTERVENTIONS:
Drug: Amantadine — Participants that have been randomized to the study group will be instructed to begin taking amantadine on the day after this study visit. They will self-administer amantadine 100 mg twice daily (morning and noon) for four weeks
  Arms: Standard of Care + Amantadine
Other: Physical, Occupational, Speech Therapy — Physical Therapy (PT) and Occupational Therapy (OT) train patients on breathing exercises and gradual reconditioning. Patients are referred to speech therapy (SLP) for cognitive remediation and metacognitive strategies.
Other: Provider Counseling — Clinic providers will provide counseling/education on Long-COVID.
Other: Medications for symptoms management — Clinic providers may recommend targeted pharmacologic management for symptoms the patient is experience. As an example, if a patient reports a headache the provider may recommend over-the-counter or prescription medications to target this particular symptom.

SUMMARY:
Purpose: To decrease symptom burden, improve cognitive function, improve endurance, and decrease fatigue in subjects with post-acute sequelae of COVID-19 (PASC) or "long-hauler" COVID using amantadine. If amantadine use is determined to be efficacious in this population, the findings of this study will be used towards a subsequent randomized control trial.

DETAILED DESCRIPTION:
This study is a prospective, open-label, single-blind, randomized control study. Study duration is approximately 6 weeks starting at the baseline visit. We will recruit 30 participants (15 per arm) for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-65
* Can provide informed consent
* Confirmed COVID+ test (either rapid antigen or PCR) between 8 weeks and one year prior to initial visit.
* Able to consent in English
* Endorse symptoms during their initial evaluation and history with the provider that began around the time of the acute COVID19 infection (subjective) including cognitive changes such as cognitive fatigue, brain fog, memory issues,attention issues AND have symptoms in at least 1 out of the 2 following symptom categories:
* Category 1: Decreased endurance, physical fatigue, weakness
* Category 2: Depression, anxiety

Exclusion Criteria:

* Known hypersensitivity to amantadine
* Clinically significant psychiatric, neurologic, renal, hepatic, opthalmologic, cardiac impairment in the opinion of the investigators, including but not limited to:
* Psychiatric:
* Acute or chronic unstable Axis I psychiatric illness
* History of psychosis
* Severe depression Patient Health Questionnaire-9 (PHQ-9) score >= 20
* Suicidality
* Neurologic:
* Epilepsy
* Cognitive dysfunction predating COVID infection
* History of delirium
* Neurologic conditions with agitation or confusion

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Measures of cognitive functioning | 4 weeks
  Repeatable Battery for the Assessment of Neuropsychological Status (R BANS) Self-reported percent back to normal, FAS, Trails A&B, and Digit
  Vigilance Test (DVT)
Measures of cognitive functioning | 4 weeks
  Cognitive Subscale of Modified Fatigue Impact Scale (MFIS)
Measures of cognitive functioning | 4 weeks
  Self-reported percent back to normal
Measures of cognitive functioning | 4 weeks
  FAS Test
Measures of cognitive functioning | 4 weeks
  Trails A & B
Measures of cognitive functioning | 4 weeks
  Digit Vigilance Test

SECONDARY OUTCOMES:
Measures of endurance and strength | 4 weeks
  6 Minute Walk Test (6MWT)
Measures of endurance and strength | 4 weeks
  30 second sit-to-stand
Measures of endurance and strength | 4 weeks
  grip strength
  grip strength
Measures of endurance and strength | 4 weeks
  Physical Function subsection of PROMIS-29
Measures of fatigue | 4 weeks
  Physical Subscale of the Modified Fatigue Impact Scale
  (MFIS), and fatigue subsection of PROMIS-29.
Measures of anxiety and depression | 4-6 weeks
  Patient Health Questionnaire-9 (PHQ-9)
Measures of anxiety and depression | 4-6 weeks
  Generalized Anxiety DIsorder-7 (GAD-7) questionnaires
Measures of anxiety and depression | 4-6 weeks
  anxiety and depression sections of the PROMIS-29

CONTACTS AND LOCATIONS:
Overall Officials: Amy Mathews, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No